CLINICAL TRIAL: NCT03868956
Title: Safety of a Management Strategy Based on Colour Doppler ULTrasound and D-Dimer Testing for the Diagnosis Exclusion of RECurrent Deep Vein Thrombosis of the Lower Limbs. The ULTREC Project
Brief Title: Diagnosis Exclusion of Recurrent Deep Vein Thrombosis of the Lower Limbs
Acronym: ULTREC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Collaborators: Centre Hospitalier Universitaire de Saint Etienne (Other); Investigation network on venous thrombo-embolism (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018-CHITS-04; 2019-A00136-51 (Other: Id-RCB)
Record Dates: First submitted 2019-03-08; First posted 2019-03-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Deep Vein Thrombosis
Keywords: Deep vein thrombosis; Recurrence; Diagnostic strategy; Colour doppler ultrasound; D-dimer
MeSH Terms: conditions — Venous Thrombosis; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic strategy (Experimental): Colour doppler ultrasound (CDUS) with or without D-dimer test to rule-in or rule-out deep vein thrombosis recurrence
  Interventions: Diagnostic Test: Colour doppler ultrasound with or without D-dimer test

INTERVENTIONS:
Diagnostic Test: Colour doppler ultrasound with or without D-dimer test — * Positive CDUS: anticoagulant treatment
  * Negative CDUS: no anticoagulant treatment
  * Non diagnostic CDUS : reference to routine D-dimer test
    * Negative test : no anticoagulant treatment
    * Positive test : second CDUS 7 days (±2) after first one
      * No change in CDUS : no anticoagulant treatment
      * Change in CDUS : anticoagulant treatment

SUMMARY:
The purpose is to assess the safety of a management strategy based on colour doppler ultrasound (CDUS) and D-Dimer test results for the diagnosis exclusion of recurrent deep vein thrombosis (DVT) of the lower limbs.

DVT recurrence requires using anticoagulant treatment to prevent thrombosis progression. Given an increased bleeding risk with prolonged treatment, an accurate diagnosis for recurrence is needed. However, the diagnosis of a new thrombosis in a previously involved leg is difficult. Imaging modalities and criteria that are currently used for the diagnosis may be equivocal and unable to discriminate between an old clot and a new one recently developed at the same site. An increase in vein diameter after vein compression by the ultrasound probe was suggested as a diagnostic criterion for a new DVT. This method has many limitations in clinical practice, mainly a lack of availability of a previous measurement and a poor inter-observer agreement.

Colour Doppler ultrasound enables to study both the thrombus and the blood flow characteristics that might help to overcome these limitations. CDUS is a well-known method for the diagnosis of vascular diseases and is used in every day clinical practice for the diagnosis of a first DVT and DVT recurrence but CDUS has never been assessed for DVT recurrence in a study. The diagnosis of DVT recurrence may be easily established using the same criteria as for a first DVT episode. Our hypothesis is that CDUS associated with D-Dimer can safely rule out the diagnosis of DVT recurrence while maintaining a good specificity.

The strategy consists in performing first a CDUS that helps to classify patients as having (positive CDUS) or not having (negative CDUS) a new thrombosis. In the case of an equivocal CDUS, a D-Dimer test is performed. If the D-dimer is normal, the diagnosis of DVT recurrence is ruled out and the patient is not treated. If the D-dimer is abnormal, the diagnosis cannot be excluded nor confirmed and a second CDUS is performed on D7±2. Meanwhile, patients are not treated by anticoagulants. An unchanged CDUS on D7±2 qualifies patients as free from a new DVT and they are not treated. Conversely a change in CDUS qualifies patients as having a new DVT which requires anticoagulant treatment.

All patients have a 3-month follow-up for the assessment of potential venous thromboembolic events.

DETAILED DESCRIPTION:
Venous thromboembolism (VTE) recurrence is a common situation after stopping anticoagulant treatment. This recurrence requires extended anticoagulant therapy to prevent thrombosis progression and embolization, but given an increased bleeding risk with prolonged treatment, an accurate diagnosis for VTE recurrence is needed.

Unfortunately, there is no reference standard for the diagnosis of deep vein thrombosis (DVT) recurrence and objective and accurate diagnostic methods are lacking. Clinical assessment does not allow discriminating between a previous and a recent thrombosis and there is no clinical prediction rule specific to the suspicion of DVT recurrence. D-dimer assays alone may not be able to safely exclude the diagnosis of DVT recurrence, and they have not been sufficiently validated in combination with clinical probability. The same holds for imaging modalities because normalisation rate after proximal DVT is low and a "residual thrombosis" may make difficult the diagnosis of a new thrombosis episode at the same site. Phlebography is non-diagnostic in 33% of cases. CT-venography has never been evaluated and MRI direct thrombus imaging (MRDTI) although very promising is still under evaluation.

As compression ultrasound (CUS) may be equivocal due to a residual thrombosis, a comparison to baseline measurements of residual vein diameter after full compression at the common femoral and the popliteal vein segments in cross-sectional plane has been suggested with an increase in diameter superior to 2 or 4 mm as a diagnosis criterion. This method has many major limitations related to: 1/the need for a previous measurement almost never available in practice, 2/ the potential for recurrence at a different site than that previously measured, 3/ a poor inter-observer agreement or at least inconsistent inter-observer variability between studies, 4/ small sample sizes in diagnostic accuracy and in diagnostic management studies and 5/ lack of external validation. Due to these limitations, recurrent ipsilateral DVT is mainly diagnosed by CUS when it occurs in a new or a normalised vein segment.

Colour Doppler ultrasound (CDUS) enables to study both the thrombus and the blood flow characteristics that might help to overcome the limitations of CUS and diameter measurements. Although CDUS has never been assessed for DVT recurrence in a study, it is used in every day clinical practice and seems very helpful. The diagnosis may be easily established using the same CDUS criteria as for a first DVT episode. Our hypothesis is that CDUS associated with D-Dimer can safely exclude the diagnosis of recurrent DVT while maintaining a good specificity.

The strategy consists in performing first a CDUS that helps to classify patients as having (positive CDUS) or not having (negative CDUS) a new thrombosis. In the case of an equivocal (non-diagnostic) CDUS, a D-Dimer test is performed followed by repeat CDUS on D7±2 if D-dimer test result is abnormal. Meanwhile, patients are not treated by anticoagulants. A negative D-dimer test or an unchanged CDUS on D7±2 qualifies patients as free from a new DVT. Conversely a change in CDUS qualifies patients as having a new DVT. Only patients with a new DVT are treated. All patients have a 3-month follow-up for the assessment of venous thromboembolic and bleeding events by an independent adjudication committee.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Known history of objectively documented deep vein thrombosis of the lower limb (with or without pulmonary embolism)
* Out-patients referred for clinically suspected acute recurrent ipsilateral DVT of the lower limb i.e. the occurrence of new symptoms and signs of DVT or the increase of symptoms and signs in patients with post-thrombotic syndrome
* Patients covered by social security or equivalent regimen
* Signed and dated informed consent

Exclusion Criteria:

* Known current pregnancy
* Any condition, which, in the opinion of the investigator may prevent him from performing the colour doppler ultrasound test (plaster cast, inaccessible vein segment after abdominal or pelvic surgery, or other causes that may lead to a technically inadequate CDUS)
* Delay from onset of symptoms to inclusion of more than 10 days
* Therapeutic anticoagulation for more than 48 hours in the two days prior to consent or a need for long term anticoagulation
* Prophylactic anticoagulation for more than 48 hours in the two days prior to consent
* Clinical symptoms of pulmonary embolism
* Life expectancy less than 3 months
* Patient unable to adhere to protocol or follow-up visits and contacts
* Participants under legal guardianship or incapacitation
* Patient already enrolled in a deep vein thrombosis (DVT) diagnostic research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 466 (Actual)
Dates: Start 2020-01-17 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Adjudicated symptomatic venous thromboembolic events | 3 months
  Rate of adjudicated symptomatic venous thromboembolic (VTE) events among patients not treated by anticoagulants according to the diagnostic strategy
  The criteria for recurrent VTE include:
  * objectively confirmed pulmonary embolism (PE) by either CT pulmonary angiography or ventilation-perfusion scan,
  * death due to PE,
  * and recurrent DVT of the leg Death, cause of death, VTE comprising isolated proximal or distal DVT and PE (with or without DVT), will be adjudicated by an independent clinical event committee blinded to the classification of the diagnostic strategy.

SECONDARY OUTCOMES:
Prevalence of deep vein thrombosis recurrence | Up to 3 months
  Proportion of patients with a new DVT among all patients included based on the results of the diagnostic tests used in the strategy and on the occurrence of VTE events during follow-up in patients untreated
Proportion of patients tested negative | A day if the diagnostic strategy is conclusive (either positive or negative) at day 0, or 7 days if it is inconclusive
  Proportion of patients tested negative by the strategy for DVT recurrence among all patients included
Proportion of complete patients | 3 months
  Proportion of patients who completed the strategy
Bleeding complication occurrence | 3 months
  The occurrence of bleeding complications will be assessed among all patients included during a 3-month follow-up period. The severity of these complications will be adjudicated by the independent clinical event committee according to the International Society on Thrombosis and Haemostasis classification criteria.
Correlation of possible strategy failure in not anticoagulated patients and patient characteristics | 3 months
  Identification of clinical and ultrasound factors which could explain failure of the strategy in non anticoagulated patients
Prevalence of isolated superficial vein thrombosis | 3 months
  Proportion of patients with isolated superficial vein thrombosis during a 3-month follow-up among all patients included

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Elias, MD, Study Director — Centre Hospitalier Intercommunal Toulon La Seyne sur Mer
Locations (45):
- France (45):
  - Centre Hospitalier de Vichy, Vichy, Allier
  - Centre Hospitalier Universitaire de Nice, Nice, Alpes-Maritimes
  - Centre Hospitalier de Carcassonne, Carcassonne, Aude
  - Centre d'angiologie, Carcassonne, Aude
  - APHM La Timone, Marseille, Bouches Du Rhône
  - Cabinet libéral Pung, Aubagne, Bouches-du-Rhône
  - Cabinet libéral Dias, Istres, Bouches-du-Rhône
  - Cabinet libéral Sidoli, Marseille, Bouches-du-Rhône
  - Cabinet libéral El Haddad, Marseille, Bouches-du-Rhône
  - Cabinet libéral De Mari, Ajaccio, Corse Du Sud
  - Cabinet libéral Secondi, Ajaccio, Corse Du Sud
  - Centre Hospitalier Universitaire Bocage, Dijon, Cote d'Or
  - Centre Hospitalier Universitaire François Mitterrand, Dijon, Côte d'Or
  - Centre hospitalier Universitaire Cavale Blanche, Brest, Finistère
  - Centre Hospitalier Universitaire de Nîmes, Nîmes, Gard
  - Centre Hospitalier d'Auch, Auch, Gers
  - Cabinet libéral Cazaux, Auch, Gers
  - Hôpital Saint André, Bordeaux, Gironde
  - Centre de medicine vasculaire interventionnel, Langon, Gironde
  - Cabinet libéral Casanova, Bastia, Haute Corse
  - Cabinet libéral Bonavita, Bastia, Haute-Corse
  - Cabinet libéral Bourrinet, Balma, Haute-Garonne
  - Centre Hospitalier Universitaire Rangueil, Toulouse, Haute-Garonne
  - Clinique Rive Gauche, Toulouse, Haute-Garonne
  - Cabinet libéral Wagner, Lourdes, Hautes-Pyrénées
  - Cabinet libéral Esteve, Tarbes, Hautes-Pyrénées
  - Centre Hospitalier Universitaire de Montpellier, Montpellier, Hérault
  - Centre Hospitalier Universitaire de Rennes, Rennes, Ille-et-Vilaine
  - Centre Hospitalier Universitaire de Grenoble, Grenoble, Isère
  - Centre Hospitalier Universitaire d'Angers, Angers, Maine-et-Loire
  - Centre Hospitalier Universitaire de Nancy, Nancy, Meurthe Et Moselle
  - Espace Artois Santé, Arras, Pas-de-Calais
  - Centre Hospitalier Universitaire Nord, Saint-Étienne-de-Montluc, Pays de la Loire Region
  - Centre Hospitalier Universitaire de Clermont-Ferrand, Clermont-Ferrand, Puy-de-Dôme
  - Hôpital Edouard Herriot, Lyon, Rhône
  - Centre Hospitalier Universitaire d'Amiens, Amiens, Somme
  - Cabinet libéral Besancon - polyclinique des Fleurs, Ollioules, Var
  - Clinique des Fleurs, Ollioules, Var
  - Cabinet libéral Richard, Sanary-sur-Mer, Var
  - Cabinet libéral Ben Sedrine, Six-Fours-les-Plages, Var
  - Cabinet libéral Riviere, Six-Fours-les-Plages, Var
  - Cabinet libéral Zimmermann, Six-Fours-les-Plages, Var
  - Centre Hospitalier Intercommunal Toulon La Seyne sur Mer, Toulon, Var
  - Hôpital Saint Joseph, Paris
  - Centre d'explorations vasculaires, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ageno W, Squizzato A, Wells PS, Buller HR, Johnson G. The diagnosis of symptomatic recurrent pulmonary embolism and deep vein thrombosis: guidance from the SSC of the ISTH. J Thromb Haemost. 2013 Aug;11(8):1597-602. doi: 10.1111/jth.12301. No abstract available. PMID 23682905
- [Background] Aguilar C, del Villar V. Combined D-dimer and clinical probability are useful for exclusion of recurrent deep venous thrombosis. Am J Hematol. 2007 Jan;82(1):41-4. doi: 10.1002/ajh.20754. PMID 16947316
- [Background] Bates SM, Jaeschke R, Stevens SM, Goodacre S, Wells PS, Stevenson MD, Kearon C, Schunemann HJ, Crowther M, Pauker SG, Makdissi R, Guyatt GH. Diagnosis of DVT: Antithrombotic Therapy and Prevention of Thrombosis, 9th ed: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines. Chest. 2012 Feb;141(2 Suppl):e351S-e418S. doi: 10.1378/chest.11-2299. PMID 22315267
- [Background] Fraser DG, Moody AR, Morgan PS, Martel AL, Davidson I. Diagnosis of lower-limb deep venous thrombosis: a prospective blinded study of magnetic resonance direct thrombus imaging. Ann Intern Med. 2002 Jan 15;136(2):89-98. doi: 10.7326/0003-4819-136-2-200201150-00006. PMID 11790060
- [Background] Geersing GJ, Zuithoff NP, Kearon C, Anderson DR, Ten Cate-Hoek AJ, Elf JL, Bates SM, Hoes AW, Kraaijenhagen RA, Oudega R, Schutgens RE, Stevens SM, Woller SC, Wells PS, Moons KG. Exclusion of deep vein thrombosis using the Wells rule in clinically important subgroups: individual patient data meta-analysis. BMJ. 2014 Mar 10;348:g1340. doi: 10.1136/bmj.g1340. PMID 24615063
- [Background] Goodacre S, Sampson F, Thomas S, van Beek E, Sutton A. Systematic review and meta-analysis of the diagnostic accuracy of ultrasonography for deep vein thrombosis. BMC Med Imaging. 2005 Oct 3;5:6. doi: 10.1186/1471-2342-5-6. PMID 16202135
- [Background] Hamadah A, Alwasaidi T, LE Gal G, Carrier M, Wells PS, Scarvelis D, Gonsalves C, Forgie M, Kovacs MJ, Rodger MA. Baseline imaging after therapy for unprovoked venous thromboembolism: a randomized controlled comparison of baseline imaging for diagnosis of suspected recurrence. J Thromb Haemost. 2011 Dec;9(12):2406-10. doi: 10.1111/j.1538-7836.2011.04533.x. PMID 21985174
- [Background] Hassen S, Barrellier MT, Seinturier C, Bosson JL, Genty C, Long A, Pernod G. High percentage of non-diagnostic compression ultrasonography results and the diagnosis of ipsilateral recurrent proximal deep vein thrombosis: a rebuttal. J Thromb Haemost. 2011 Feb;9(2):414-6; author reply 417-8. doi: 10.1111/j.1538-7836.2010.04137.x. No abstract available. PMID 21070594
- [Background] Heijboer H, Jongbloets LM, Buller HR, Lensing AW, ten Cate JW. Clinical utility of real-time compression ultrasonography for diagnostic management of patients with recurrent venous thrombosis. Acta Radiol. 1992 Jul;33(4):297-300. PMID 1633039
- [Background] Hull RD, Carter CJ, Jay RM, Ockelford PA, Hirsch J, Turpie AG, Zielinsky A, Gent M, Powers PJ. The diagnosis of acute, recurrent, deep-vein thrombosis: a diagnostic challenge. Circulation. 1983 Apr;67(4):901-6. doi: 10.1161/01.cir.67.4.901. PMID 6825247
- [Background] Kearon C, Akl EA, Ornelas J, Blaivas A, Jimenez D, Bounameaux H, Huisman M, King CS, Morris TA, Sood N, Stevens SM, Vintch JRE, Wells P, Woller SC, Moores L. Antithrombotic Therapy for VTE Disease: CHEST Guideline and Expert Panel Report. Chest. 2016 Feb;149(2):315-352. doi: 10.1016/j.chest.2015.11.026. Epub 2016 Jan 7. PMID 26867832
- [Background] Le Gal G, Righini M, Roy PM, Sanchez O, Aujesky D, Perrier A, Bounameaux H. Value of D-dimer testing for the exclusion of pulmonary embolism in patients with previous venous thromboembolism. Arch Intern Med. 2006 Jan 23;166(2):176-80. doi: 10.1001/archinte.166.2.176. PMID 16432085
- [Background] Le Gal G, Kovacs MJ, Carrier M, Do K, Kahn SR, Wells PS, Anderson DA, Chagnon I, Solymoss S, Crowther M, Righini M, Perrier A, White RH, Vickars L, Rodger M. Validation of a diagnostic approach to exclude recurrent venous thromboembolism. J Thromb Haemost. 2009 May;7(5):752-9. doi: 10.1111/j.1538-7836.2009.03324.x. Epub 2009 Feb 18. PMID 19228281
- [Background] Linkins LA, Stretton R, Probyn L, Kearon C. Interobserver agreement on ultrasound measurements of residual vein diameter, thrombus echogenicity and Doppler venous flow in patients with previous venous thrombosis. Thromb Res. 2006;117(3):241-7. doi: 10.1016/j.thromres.2005.02.011. Epub 2005 Mar 21. PMID 16378830
- [Background] Prandoni P, Cogo A, Bernardi E, Villalta S, Polistena P, Simioni P, Noventa F, Benedetti L, Girolami A. A simple ultrasound approach for detection of recurrent proximal-vein thrombosis. Circulation. 1993 Oct;88(4 Pt 1):1730-5. doi: 10.1161/01.cir.88.4.1730. PMID 8403319
- [Background] Prandoni P, Lensing AW, Bernardi E, Villalta S, Bagatella P, Girolami A; DERECUS Investigators Group. The diagnostic value of compression ultrasonography in patients with suspected recurrent deep vein thrombosis. Thromb Haemost. 2002 Sep;88(3):402-6. PMID 12353067
- [Background] Prandoni P, Tormene D, Dalla Valle F, Concolato A, Pesavento R. D-dimer as an adjunct to compression ultrasonography in patients with suspected recurrent deep vein thrombosis. J Thromb Haemost. 2007 May;5(5):1076-7. doi: 10.1111/j.1538-7836.2007.02455.x. Epub 2007 Mar 15. No abstract available. PMID 17367489
- [Background] Rathbun SW, Whitsett TL, Raskob GE. Negative D-dimer result to exclude recurrent deep venous thrombosis: a management trial. Ann Intern Med. 2004 Dec 7;141(11):839-45. doi: 10.7326/0003-4819-141-11-200412070-00007. PMID 15583225
- [Background] Schulman S, Granqvist S, Holmstrom M, Carlsson A, Lindmarker P, Nicol P, Eklund SG, Nordlander S, Larfars G, Leijd B, Linder O, Loogna E. The duration of oral anticoagulant therapy after a second episode of venous thromboembolism. The Duration of Anticoagulation Trial Study Group. N Engl J Med. 1997 Feb 6;336(6):393-8. doi: 10.1056/NEJM199702063360601. PMID 9010144
- [Background] Tan M, Velthuis SI, Westerbeek RE, VAN Rooden CJ, VAN DER Meer FJ, Huisman MV. High percentage of non-diagnostic compression ultrasonography results and the diagnosis of ipsilateral recurrent proximal deep vein thrombosis. J Thromb Haemost. 2010 Apr;8(4):848-50. doi: 10.1111/j.1538-7836.2010.03758.x. No abstract available. PMID 20398187
- [Background] Tan M, Bornais C, Rodger M. Interobserver reliability of compression ultrasound for residual thrombosis after first unprovoked deep vein thrombosis. J Thromb Haemost. 2012 Sep;10(9):1775-82. doi: 10.1111/j.1538-7836.2012.04827.x. PMID 22726359
- [Background] Tan M, Mol GC, van Rooden CJ, Klok FA, Westerbeek RE, Iglesias Del Sol A, van de Ree MA, de Roos A, Huisman MV. Magnetic resonance direct thrombus imaging differentiates acute recurrent ipsilateral deep vein thrombosis from residual thrombosis. Blood. 2014 Jul 24;124(4):623-7. doi: 10.1182/blood-2014-04-566380. Epub 2014 Jun 13. PMID 24928859
- [Background] van der Hulle T, Tan M, den Exter PL, van Roosmalen MJ, van der Meer FJ, Eikenboom J, Huisman MV, Klok FA. Recurrence risk after anticoagulant treatment of limited duration for late, second venous thromboembolism. Haematologica. 2015 Feb;100(2):188-93. doi: 10.3324/haematol.2014.112896. Epub 2014 Sep 26. PMID 25261098
- [Background] Westerbeek RE, Van Rooden CJ, Tan M, Van Gils AP, Kok S, De Bats MJ, De Roos A, Huisman MV. Magnetic resonance direct thrombus imaging of the evolution of acute deep vein thrombosis of the leg. J Thromb Haemost. 2008 Jul;6(7):1087-92. doi: 10.1111/j.1538-7836.2008.02986.x. Epub 2008 Jul 1. PMID 18433464